CLINICAL TRIAL: NCT06083155
Title: The NetherLands Registry of Invasive Coronary Vasomotor Function Testing (NL-CFT)
Acronym: NL-CFT
Status: Enrolling by invitation | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Catharina Ziekenhuis Eindhoven (Other); Maasstad Hospital (Other); VieCuri Medical Centre (Other); Frisius Medisch Centrum (Other); Haaglanden Medical Centre (Other); Rijnstate Hospital (Other); Medisch Spectrum Twente (Other); Onze Lieve Vrouwe Gasthuis (Other); Tergooi Hospital (Other); Amphia Hospital (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Noordwest Ziekenhuisgroep (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 79233
Record Dates: First submitted 2023-08-23; First posted 2023-10-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Coronary Vasospasm; Coronary Microvascular Dysfunction; Non-Obstructive Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Vasospasm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal CFT results: no coronary vasomotor dysfunction: Collection of data on anginal complaints, use of medication and major adverse cardiac events (MACE) by means of online patient questionnaires
  Interventions: Diagnostic Test: Coronary Function Test; Other: Patient questionnaires
- Abnormal CFT results: coronary vasomotor dysfunction: Comparison of patient reported outcomes of different endotype groups Collection of data on anginal complaints, use of medication and MACE by means of online patient questionnaires
  Interventions: Diagnostic Test: Coronary Function Test; Other: Patient questionnaires

INTERVENTIONS:
Diagnostic Test: Coronary Function Test — All participants are referred for a clinically indicated coronary function test
Other: Patient questionnaires — All participants that consent will receive yearly followup questionnaires for 5 years after their initial consent

SUMMARY:
The goal of this registry is to collect data on patients referred for clinically indicated coronary vasomotor function test (CFT) and answer different questions on prevalence, safety and outcomes. The registry is observational. Patients receive yearly online questionnaires on their anginal complaints for 5 years after their CFT.

ELIGIBILITY:
Inclusion Criteria:

* Referred for clinically indicated CFT

Exclusion Criteria:

* Not willing to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred for clinically indicated CFT are eligible
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of coronary vasomotor dysfunction | Baseline
  Can be handled as dichotomous outcome with normal vs abnormal coronary function test (CFT) results. Alternatively, can also be handled as categorical outcome with the following categories.
  1. Normal CFT results
  2. Vasospastic endotype (epicardial or microvascular); tested by acetylcholine provocation
  3. Microvascular dysfunction endotype (decreased coronary flow reserve or increased index of microvascular resistance); tested by bolus thermodilution, optionallly with additional continuous thermodilution method
  4. Mixed endotype

SECONDARY OUTCOMES:
Angina burden | Baseline and every year up to 5 years after baseline
  Measured by Seattle Angina Questionnaire summary score, 0-100 with higher scores indicating better (functional) status.
Experienced quality of life | Baseline and every year up to 5 years after baseline
  Measured by Short Form 36, 0-100 with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter Damman, Principal Investigator — Radboud University Medical Center
Locations (15):
- Netherlands (15):
  - RadboudUMC, Nijmegen, Gelderland
  - Amsterdam UMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Tergooi Hospital, Hilversum
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maastricht UMC, Maastricht
  - Maasstad Ziekenhuis, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - Elisabeth-TweeSteden Hospital, Tilburg
  - UMC Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: No
Only participating centers that signed the joint data registry agreement can make a request for data after approval of steering committee.

REFERENCES:
- [Derived] Crooijmans C, Jansen TPJ, Meeder JG, Paradies V, de Vos AMJ, Woudstra P, Vossenberg TNE, van de Hoef TP, Vos NS, Olde Bijvank EGM, van den Oord SCH, Winkler P, Meuwissen M, Widdershoven JWMG, Arkenbout EK, Stoel MG, Appelman Y, Beijk MAM, Cetinyurek-Yavuz A, den Ruijter HM, Elias-Smale SE, van Royen N, Dimitriu-Leen AC, Damman P; for NL-CFT. Angina Severity and Symptom Improvement Are Associated With Diagnostic Acetylcholine Provocation Dose in Vasospastic Angina. J Am Heart Assoc. 2025 Jan 21;14(2):e037913. doi: 10.1161/JAHA.124.037913. Epub 2025 Jan 16. PMID 39818972